CLINICAL TRIAL: NCT06054919
Title: The Effect of Vitamin D3 Therapy on 25(OH)D, 1,25(OH)2D, VDBP, and 24,25(OH)2D Maternal Serum Levels in Pregnant Women With Vitamin D Deficient and Insufficient
Brief Title: The Effect of Vitamin D3 Therapy on Vitamin D Status in Pregnant Women With Vitamin D Deficient and Insufficient
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Rima Irwinda, MD, OBGYN, PhD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 257/UN.2F1/ETIK/PPM.00.02/2023
Record Dates: First submitted 2023-09-05; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50,000 IU (Experimental): Vitamin D3 50,000 IU weekly a standard prenatal multivitamin (fumarate Fe 90 mg; folic acid 0.4 mg; vitamin B6 3 mg; vitamin B12 5 mcg; sulphate cupric 0.35 mg, sulphate cobalt 0.15 mg, sulphate mangan 5 mcg, vitamin C 60 mg, vitamin E 5 mg, and phosphate calcium 60 mg)
  Interventions: Drug: Cholecalciferol
- 5,000 IU (Active Comparator): Vitamin D3 5,000 IU daily a standard prenatal multivitamin (fumarate Fe 90 mg; folic acid 0.4 mg; vitamin B6 3 mg; vitamin B12 5 mcg; sulphate cupric 0.35 mg, sulphate cobalt 0.15 mg, sulphate mangan 5 mcg, vitamin C 60 mg, vitamin E 5 mg, and phosphate calcium 60 mg)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — vitamin D3
  Other Names: vitamin D

SUMMARY:
This study is a randomized controlled trial which compares the effect of vitamin D3 therapy 5,000 IU daily and 50,000 IU on 25(OH)D and 1,25(OH)2D, VDBP, and 24,25(OH)2D maternal serum levels in pregnant women with vitamin D deficient and insufficient.

DETAILED DESCRIPTION:
This is a randomized controlled trial of vitamin D therapy of 5,000 IU daily or 50,000 IU weekly during pregnancy. The study is conducted at Cipto Mangunkusumo National Center General Hospital and Koja Distict Hospital in Jakarta, Indonesia from April 2021 - December 2023. All the pregnant women are screened for eligibility when they presented to the clinic for antenatal care visits and are offered enrolment if they meet the following inclusion criteria: gestational age of ≤ 14 weeks, vitamin D deficient or insufficient (25(OH)D <30 ng/ml], and positive fetal heart rate from ultrasound examination.

Participants are randomly assigned to one of two parallel intervention groups, with allocation concealment: vitamin D3 (cholecalciferol) 5,000 IU/week or 50,000 IU/week. All participants are given a standard prenatal multivitamin. A medical history, physical, and ultrasound examination are performed. Participants complete a questionnaire about sunlight exposure. Interventions in both groups are given for four weeks. Baseline blood tests, including serum 25(OH)D, 1,25(OH)2D, VDBP, and 24,25(OH)2D are performed at recruitment. After four weeks of interventions, the maternal venous blood is collected to assess serum 25(OH)D, 1,25(OH)2D, VDBP, and 24,25(OH)2D.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with gestational age of ≤ 14 weeks
* vitamin D deficient or insufficient (25(OH)D <30 ng/ml]
* positive fetal heart rate from ultrasound examination.

Exclusion Criteria:

* multiple pregnancy
* pregnancy with congenital anomaly
* hyperemesis gravidarum, diarrhea
* complicated medical history (hypertension, diabetes mellitus, heart, kidney, or liver disease)
* use of any dietary supplement containing vitamin D prior to enrolment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
25(OH)D maternal serum level | 4 weeks after intervention
  quantified by direct competitive Chemilumiscence Immunoassay (CLIA) using LIAISON®.
1,25(OH)2D maternal serum level | 4 weeks after intervention
  quantified by Liquid Chromatography-tandem Mass Spectrometry (LC-MS/MS) using ImmuTube®.
VDBP maternal serum level | 4 weeks after intervention
  quantified by Enzyme-Linked Immunosorbent Assay (ELISA) using Quantikine®
24,25(OH)2D maternal serum level | 4 weeks after intervention
  quantified by Acquity I Class Binary Solvent Manager FTN , Xevo TQXS Tandem Mass Spectrometry (Waters Corporation)

CONTACTS AND LOCATIONS:
Overall Officials: Rima Irwinda, MD, PhD, Study Chair — Departement of Obstetrics and Gynecology, Faculty of Medicine University of Indonesia
Locations (1):
- Cipto Mangunkusumo National Center General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
The research findings will be disseminated via publication of results, submission of information to public accessible databases, or meetings
Supporting Information: Study Protocol
Time Frame: the data will become available in June 2024
Access Criteria: there is no access criteria

REFERENCES:
- [Derived] Syafitri I, Irwinda R, Saroyo YB, Purwosunu Y, Wibowo N. Maternal concentrations of vitamin D metabolites in response to high-dose oral vitamin D during first trimester pregnancy: a randomized controlled trial. BMC Nutr. 2025 Jul 4;11(1):117. doi: 10.1186/s40795-025-01104-3. PMID 40616177

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT06054919/Prot_SAP_000.pdf